CLINICAL TRIAL: NCT04605731
Title: A Phase Ib Study of Durvalumab (Medi4736) and Tremelimumab Following Radioembolization in Patients With Unresectable Locally Advanced Hepatocellular Carcinoma
Brief Title: Durvalumab and Tremelimumab After Radioembolization for the Treatment of Unresectable, Locally Advanced Liver Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20187; NCI-2020-06932 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20187 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: BCLC Stage B Hepatocellular Carcinoma; BCLC Stage C Hepatocellular Carcinoma; Locally Advanced Hepatocellular Carcinoma; Stage III Hepatocellular Carcinoma AJCC v8; Stage IIIA Hepatocellular Carcinoma AJCC v8; Stage IIIB Hepatocellular Carcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IVA Hepatocellular Carcinoma AJCC v8; Stage IVB Hepatocellular Carcinoma AJCC v8; Unresectable Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab; Immunoglobulin G; Disulfides; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (durvalumab, tremelimumab) (Experimental): Patients undergo standard of care radioembolization with Yttrium-90 SIR-spheres intra-arterially over 60-90 minutes on day -14. Patients then receive durvalumab IV over 1 hour and tremelimumab IV over 1 hour on day 1. Cycles with durvalumab repeat every 4 weeks for 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Biological: Tremelimumab

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Ticilimumab

SUMMARY:
This phase Ib trial investigates the side effects of durvalumab and tremelimumab after radioembolization (radiation particles against liver tumors) and to see how well they work in treating patients with liver cancer that cannot be removed by surgery (unresectable) and has spread to nearby tissues and lymph nodes (locally advanced). Durvalumab and tremelimumab are antibodies (proteins produced by the defense system of the body [immune system]) that have been made in the laboratory and may improve the ability of the immune system to detect and fight cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the safety of durvalumab and tremelimumab following radioembolization with Yttrium-90 selective internal radiation (SIR)-spheres in patients with locally advanced hepatocellular carcinoma without extra-hepatic disease.

II. If the combination of durvalumab and tremelimumab is deemed unsafe, to establish the safety of single agent durvalumab and explore all endpoints with durvalumab alone.

III. To evaluate the overall response rate in patients treated with durvalumab and tremelimumab following radioembolization with Yttrium-90 SIR-Spheres using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, modified (m) RECIST and immune modified RECIST criteria.

SECONDARY OBJECTIVES:

I. To evaluate the rate of 6-month progression-free survival in patients treated with durvalumab and tremelimumab following radioembolization with Yttrium-90 SIR-spheres.

II. To evaluate median progression-free survival and overall survival in patients treated with durvalumab and tremelimumab following radioembolization with Yttrium-90 SIR-spheres.

EXPLORATORY OBJECTIVES:

I. To explore the association of response and survival outcomes with PD-L1 expression of baseline tumor biopsies.

II. To explore the association of response and survival outcomes with next generation sequencing results including tumor mutational burden of baseline tumor biopsies.

III. To explore genomic alterations/evolutions in tumor tissue following Yttrium-90 SIR-spheres and durvalumab plus tremelimumab through comparison of baseline and post-combination immunotherapy treatment tumor biopsies.

IV. To explore the association of response and survival outcomes with gene expression signatures.

OUTLINE:

Patients undergo standard of care radioembolization with Yttrium-90 SIR-spheres intra-arterially over 60-90 minutes on day -14. Patients then receive durvalumab intravenously (IV) over 1 hour and tremelimumab IV over 1 hour on day 1. Cycles with durvalumab repeat every 4 weeks for 12 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 90 days, and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed unresectable, locally advanced hepatocellular carcinoma as defined by Barcelona Clinic Liver Cancer (BCLC) (B) intermediate stage or BCLC (C) advanced stage without extra-hepatic disease (only with branch portal vein thrombosis)
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act in the United States [US]) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Must have a life expectancy of at least 12 weeks
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
* Male patients must be surgically sterile, or if sexually active and having a pre-menopausal female partner then must be using an acceptable form of contraception
* Have a Child-Pugh class A liver score within 7 days of radioembolization
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as outlined in RECIST version 1.1
* Patients should have been identified by their respective physicians as candidates for radioembolization
* Body weight > 30 kg
* Subjects with chronic infection by hepatitis C virus (HCV) who are untreated are allowed on study. In addition, subjects with successful HCV treatment (defined as sustained virologic response [SVR] 12 or SVR 24) are allowed as long as 4 weeks have passed between completion of HCV therapy and start of study drug
* Subjects with hepatitis B virus (HBV) may only be enrolled if their hepatitis is judged clinically stable by the investigator
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelet count >= 75000/uL
* Total bilirubin < 2.0 mg/dL. This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician
* Aspartate aminotransferase (AST/serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT/serum glutamate pyruvate transaminase [SGPT]) =< 5 x upper limit of normal (ULN)
* Albumin >= 2.8 g/dL
* International normalized ration =< 1.6
* Measured creatinine clearance (CL) > 40 mL/min or calculated creatinine CL > 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance

Exclusion Criteria:

* Portal vein invasion at the main portal branch (Vp4), inferior vena cava, or cardiac involvement of hepatocellular carcinoma (HCC) based on imaging. Vascular invasion to portal vein side branches are eligible for study
* Evidence of diffuse HCC (tumor burden occupying > 50% of liver)
* Any evidence of known metastatic disease
* Major surgical procedure (as defined by the investigator) within 28 days prior to radioembolization

  * Note: Local surgery of isolated lesions for palliative intent is acceptable
* Participation in another clinical study with an investigational product during the last 4 weeks
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) =< 28 days prior to the first dose of study drug. If sufficient wash-out time has not occurred due to the schedule or pharmacokinetic (PK) properties of an agent, a longer wash-out period will be required, as agreed by AstraZeneca/MedImmune and the investigator
* Prior exposure to anti-PD-1/PD-L1 inhibitor or anti-CTLA4 inhibitor, including durvalumab or tremelimumab
* Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade >= 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
* Patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab and/or tremelimumab may be included only after consultation with the study physician
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* History of allogenic organ transplantation
* Evidence of pulmonary lung shunt greater than 10% or expected lung dose of > 30 Gy
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent
* History of another primary malignancy except for

  * Malignancy treated with curative intent and with no known active disease >= 5 years before the first dose of study treatment and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* History of active primary immunodeficiency
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study treatment

  * Note: Patients, if enrolled, should not receive live vaccine whilst receiving study treatment and up to 30 days after the last dose of study treatment
* Active systemic infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis (TB) testing in line with local practice. Use of antibiotics to treat superficial infection or contamination of tumor shall not, by itself, be considered evidence of infection
* History of leptomeningeal carcinomatosis
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
* Any concurrent chemotherapy, investigational product (IP), biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroid or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication)
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is longer
* Female subjects, unless postmenopausal or surgically sterile, unwillingness to practice effective contraception, as per investigator discretion during the study. The rhythm method is not to be used as the sole method of contraception
* Male subjects, unwillingness to practice effective contraception (per investigator discretion) while taking part in this study, because the effects of the SIR-Spheres treatment on sperm or upon the development of an unborn child are unknown
* Inability or unwillingness to understand or sign a written informed consent document
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 90 days post-last dose of durvalumab
  Will be assessed per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Dose-limiting toxicity | From the time of first administration of durvalumab or tremelimumab until 4 weeks (one cycle) after the first administration
  Will be assessed per NCI CTCAE version 5.0.
Overall response | From the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started), assessed up to 2 years
  Will be evaluated using the new updated international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) committee version 1.1, modified RECIST (mRECIST), and immune modified RECIST (imRECIST) criteria.

SECONDARY OUTCOMES:
Progression-free survival | From study enrollment to when objective evidence of disease progression is documented, assessed at 6 months
  Will be evaluated using the new updated international criteria proposed by the RECIST committee version 1.1, mRECIST, and imRECIST criteria.
Median progression-free survival | Up to 2 years
  Will be evaluated using the new updated international criteria proposed by the RECIST committee version 1.1, mRECIST, and imRECIST criteria.
Overall survival | From study enrollment until death, assessed up to 2 years

OTHER OUTCOMES:
PD-L1 expression in baseline tumor biopsies | Up to 2 years
  Will be associated with response and survival outcomes.
Tumor mutational burden | Up to 2 years
  Next generation sequencing results, including tumor mutational burden in baseline tumor biopsies, will be associated with response and survival outcomes.
Genomic alterations/evolutions | Up to 2 years
Gene expression signatures | Up to 2 years
  Will be associated with response and survival outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Daneng Li, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States